CLINICAL TRIAL: NCT03669172
Title: Fase I/II, Unicentric, Historical Control Clinical Trial to Evaluate the Effectiveness of Donor IL-15 Stimulated NK Cells Post Transplant Infusion, in Acute Leukemia Patients With Poor Prognosis and Haploidentical Unmanipulated Transplant
Brief Title: Efectiveness of Donor IL-15-stimulated NK Cells Post Transplant Infusion in in Acute Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Martín, José Luis Díez, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-HEM-HGUGM-2016-01
Record Dates: First submitted 2018-03-06; First posted 2018-09-13 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: ACUTE LEUKEMIA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK cells infusion (Experimental): NK cells incubated infusion (CD56 +, CD3) ex vivo with IL-15 in patients with acute myeloid leukemia undergoing high-risk allogeneic haploidentical Pt-C donor
  Interventions: Biological: Donor IL-15 stimulated NK cells infusion

INTERVENTIONS:
Biological: Donor IL-15 stimulated NK cells infusion — DONOR IL-15-STIMULATED NK CELLS POST TRANSPLANT INFUSION, IN ACUTE LEUKEMIA PATIENTS WITH POOR PROGNOSIS AND HAPLOIDENTICAL UNMANIPULATED TRANSPLANT

SUMMARY:
Clinical trial phase I and II, single-center, historical control, to evaluate the effectiveness of donor IL-15 stimulated NK cells post transplant infusion, in acute leukemia patients with poor prognosis and haploidentical unmanipulated transplant

DETAILED DESCRIPTION:
This clinical trial wants to study the safety, effectiveness and efficacy of NK cells incubated infusion (CD56 +, CD3) incubated ex vivo with IL-15 infusion in patients with high risk acute myeloid leukemia undergoing allogeneic transplant of an haploidentical donor with post-transplant cyclophosphamide administration.

ELIGIBILITY:
Inclusion Criteria:

1. More than 18 years old, with acute myeloid leukemia who goes to undergo haploidentical
2. Assessable disease by analytic, molecular or image techniques.
3. Comorbidity Sorror index less than 6.
4. Give informed consent according to the legal requirements.
5. Dispose of a donor without exclusion criteria.

Exclusion Criteria:

1. Positive HIV serology.
2. Patients with an active infection or other underlying serious medical statement.
3. Any medical process, analytical abnormality or important psychiatric disorder, according to the investigator's opinion, that prevent the participation of the patient in the study.
4. Participation of any other interventional clincal trial within 30 days of planned enrollment into this study.
5. Women who are pregnant or breastfeeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Up to 2 years after first infusion
  Number of Treatment-Related Adverse Events as Assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Reevaluation of the Minimal residual disease (MRD) | Up to 1 year after first infusion
  Reevaluation of the Minimal residual disease (MRD) in bone marrow by flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided